CLINICAL TRIAL: NCT05241158
Title: State Anxiety Level in Patients Undergoing Upper Gastrointestinal Endoscopy
Brief Title: Impact of Counselling and Visual Aid on Anxiety in Endoscopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, ali asad, Principle investigator, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 179/RC/KEMU
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Chronic Liver Disease; Inflammatory Bowel Diseases
Keywords: Endoscopy; Visual Aid; Anxiety; Counselling
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anxiety Disorders | interventions — Counseling; Audiovisual Aids

STUDY DESIGN:
Intervention Model Description: The patients were then randomly allocated between two groups (group 1 watched animated video of endoscopy procedure, however, group 2 didn't watch any video) on a 1:1 ratio using permuted block randomization with a fixed block sizes of four, by a house officer who wasn't involved in providing intervention to any group or in assisting any of the endoscopy procedures. The allocation sequence to the study conditions was kept concealed from psychologists measuring outcome variables, using sequentially numbered, opaque and sealed envelopes.
Who Masked: Outcomes Assessor
Masking Description: The randomisation process was performed by a house officer who was not involved in performing any of the endoscopy procedures and was responsible to break the code in case of adverse event. The allocation sequence to the study conditions was kept concealed from psychologists measuring outcome variables, using sequentially numbered, opaque and sealed envelopes. Patients were told not to inform anyone about their allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: Counselling group Patients were given a briefing about the procedure; the use of local anesthetic along with potential benefits and side effects of the drug. The steps of the endoscopy procedure (gastroscopy or colonoscopy) were explained in detail including the position, intubation, biopsy or intervention wherever applicable, extubation and post-procedure observation period in the recovery room. Detailed instructions were provided regarding post-procedural care, introduction of diet & follow-up.
  Interventions: Behavioral: Counselling
- Group B (Active Comparator): Group B: Video group Patients in the visual aid group (video group) were provided with the same information mentioned in intervention group A. In addition to that, patients watched a 5 minutes video of the respective procedure. Video showed the animation of a gastroscopy or colonoscopy procedure with a voice over explaining all the steps of the procedure in addition to the pre and post-procedure precautions to be observed.
  Interventions: Behavioral: Counselling with visual aid

INTERVENTIONS:
Behavioral: Counselling with visual aid — patients were counselled about the procedure, complications and the post-procedure recovery phase and shown a 5 minutes animated video of the gastroscopy or colonoscopy procedure
  Arms: Group B
Behavioral: Counselling — Patients counselled about the procedure, complications and the post-procedure recovery phase
  Arms: Group A

SUMMARY:
A single blind randomized controlled trial was conducted to compare the effect of counselling and visual aid on the anxiety levels in patients undergoing endoscopy and to investigate the superiority of visual aid over psychological counselling and preparation for the procedure in an informed patient.

DETAILED DESCRIPTION:
A single blind RCT was conducted to assess level of state anxiety between two interventional groups; counselling group and video group. 232 consecutive patients were enrolled from the outpatient department who were scheduled to undergo either a gastroscopy or a colonoscopy (diagnostic or therapeutic). The patients were randomly allocated to one of the two intervention groups (A and B) at the time of endoscopy scheduling. All of the patients received regular instructions regarding gut-preparation at the time of appointment and were also provided with written clear instructions. A gastroenterologist provided information about endoscopy, including the exact preparation instructions and information on the importance of bowel preparation and the adverse effects of the agents used.

Depression Anxiety Stress Scale-42 was administered at baseline. Intervention group A (counselling group) was counselled about the procedure, complications and the post-procedure recovery phase and Group B (video group) was also counselled and shown a 5 minutes animated video of the respective procedure in separate room by gastroenterologist. Endoscopies were carried out by trained doctors (endoscopists) with a minimum experience of 1000 endoscopic procedures. Patients in both the groups were interviewed again after the intervention using Depression Anxiety Stress Scale-42.

ELIGIBILITY:
Inclusion Criteria:

* both genders (male or female) with a minimum age of 18 years
* Able to comprehend questions being asked in Urdu language
* Mentally competent at signing the consent form

Exclusion Criteria:

* Patients who were diagnosed cases of psychiatric illnesses
* Undergoing emergency endoscopy (whether diagnostic or therapeutic)
* End stage renal disease
* Hearing difficulty
* Senile dementia
* Pregnant or diagnosed cases of malignancy
* Signs of hepatic encephalopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Anxiety | 90 minutes
  Depression Anxiety Stress Scale-42 (DASS-42) was used to measure state anxiety of the patients undergoing endoscopy before and after intervention.. Score on anxiety scale ranges from 0 to 20+. 0-7 is normal, 8-9 is mild, 10-14 is moderate, 15-19 is severe and 20+ is extremely severe anxiety. The higher score on anxiety scale, the higher the level of anxiety among participants.

SECONDARY OUTCOMES:
fear | 90 minutes
  Visual analogue scale was used to measure fear of the patients undergoing endoscopy before and after intervention. Participants were asked to rate the intensity of fear on a scale of 0-10. 0 means no fear and 10 means worst fear possible.
Stress | 90 minutes
  Depression Anxiety Stress Scale-42 (DASS-42) was used to measure stress of the patients undergoing endoscopy before and after intervention. Score on stress scale ranges from 0 to 34+. 0-14 is normal, 15-18 is mild, 19-25 is moderate, 26-33 is severe and 34+ is extremely severe stress. The higher score on stress scale, the higher the level of stress among participants.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asad Khan, FCPS, Principal Investigator — King Edward Medical University; Anam Ali, MS, Principal Investigator — University of Child Health Sciences & The Children's Hospital, Lahore
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan AA, Ali A, Khan AS, Shafi Y, Masud M, Irfan F, Abaidullah S. Effects of visual aid on state anxiety, fear and stress level in patients undergoing endoscopy: a randomized controlled trial. Ann Med. 2023 Dec;55(1):1234-1243. doi: 10.1080/07853890.2023.2191000. PMID 37078544